CLINICAL TRIAL: NCT07155525
Title: Pancreaticojejunostomy With or Without Modified N-butyl-2-cyanoacrylate Following Pancreaticoduodenectomy in Soft Pancreas: Randomized Controlled Trial
Brief Title: Tissue Adhesive Glue Modified Cyanoacrylate (Glubran® 2) in Soft Pancreas
Acronym: NBCA-MS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1319/10/2024
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer; Periampullary Cancer; Duodenal Cancer; Cholangiocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Head Mass; Bile Duct Cancer
Keywords: Pancreaticoduodenectomy; Pancreaticojejunostomy; Postoperative Pancreatic Fistula; Soft Pancreas; N-Butyl-2-Cyanoacrylate; Whipple procedure; Tissue adhesive; POPF prevention
MeSH Terms: conditions — Pancreatic Neoplasms; Duodenal Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Pancreaticojejunostomy; Tissue Adhesives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The operating surgeon and patient cannot be blinded due to the nature of the intervention. However, outcome assessors, including radiologists reviewing imaging studies and physicians evaluating postoperative complications, will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pancreaticojejunostomy with Modified N-Butyl-2-Cyanoacrylate (Glubran® 2) (Experimental): Patients undergo standard duct-to-mucosa pancreaticojejunostomy with topical application of 1-2 mL modified N-butyl-2-cyanoacrylate to the anastomotic site and surrounding pancreatic parenchyma.
  Interventions: Drug: Pancreaticojejunostomy with Modified N-Butyl-2-Cyanoacrylate (Glubran® 2)
- Standard Pancreaticojejunostomy without tissue adhesive application. (Active Comparator): Patients undergo duct-to-mucosa pancreaticojejunostomy without additional adhesive following pancreaticoduodenectomy.
  Interventions: Procedure: Standard(duct-to-mucosa) Pancreaticojejunostomy

INTERVENTIONS:
Drug: Pancreaticojejunostomy with Modified N-Butyl-2-Cyanoacrylate (Glubran® 2) — * Standard duct-to-mucosa pancreaticojejunostomy performed
  * Application of 0.5-1.0 mL modified N-butyl-2-cyanoacrylate around the anastomotic site
  * Adhesive applied circumferentially around the pancreaticojejunal anastomosis
  * Allow 2-3 minutes for polymerization before proceeding
  * Standard placement of peritoneal drains
  Other Names: Tissue Adhesive, Cyanoacrylate Glue,Glubran® 2
  Arms: Pancreaticojejunostomy with Modified N-Butyl-2-Cyanoacrylate (Glubran® 2)
Procedure: Standard(duct-to-mucosa) Pancreaticojejunostomy — * Patients undergo duct-to-mucosa pancreaticojejunostomy without additional adhesive following pancreaticoduodenectomy.
  * Standard placement of peritoneal drains
  * All other aspects of surgical care identical to experimental arm
  Other Names: Standard Pancreaticojejunostomy
  Arms: Standard Pancreaticojejunostomy without tissue adhesive application.

SUMMARY:
This is a single-center, randomized controlled trial comparing the efficacy of pancreaticojejunostomy with modified N-butyl-2-cyanoacrylate(Glubran® 2) versus standard pancreaticojejunostomy without cyanoacrylate in preventing postoperative pancreatic fistula (POPF) in patients undergoing pancreaticoduodenectomy with soft pancreatic texture. The primary endpoint is the incidence of postoperative pancreatic fistula at 30 days post-surgery, as defined by the International Study Group on Pancreatic Fistula (ISGPF) criteria.Secondary outcomes include surgical complications and length of hospital stay. The study will enroll approximately 194 patients at a single center.

DETAILED DESCRIPTION:
Postoperative pancreatic fistula (POPF) remains the most common and serious complication following pancreaticoduodenectomy, with incidence rates reaching up to 56.7% in patients with soft pancreatic texture. The soft pancreatic parenchyma is particularly vulnerable to anastomotic breakdown due to its friable nature and difficulty in achieving secure suturing.

N-butyl-2-cyanoacrylate is a biodegradable tissue adhesive that polymerizes rapidly upon contact with hydroxide ions in tissue fluids, forming a strong, flexible bond. The application of modified N-butyl-2-cyanoacrylate to pancreaticoenteric anastomoses may reduce the incidence of POPF by providing additional mechanical reinforcement and sealing of minor leaks.

This is a phase III, single-center, prospective, randomized controlled trial with parallel groups. Eligible patients will undergo intraoperative assessment of pancreatic texture (soft confirmed by surgeon's palpation). Randomization will occur intraoperatively after resection but before reconstruction, using computer-generated blocks.

This study aims to evaluate whether the application of modified N-butyl-2-cyanoacrylate (Glubran® 2) during pancreaticojejunostomy can significantly reduce the incidence of POPF in patients with soft pancreatic texture undergoing pancreaticoduodenectomy. Patients will be randomized to receive either standard pancreaticojejunostomy (control group) or pancreaticojejunostomy with modified N-butyl-2-cyanoacrylate application (intervention group).

The intervention group will receive 1-2 mL of modified N-butyl-2-cyanoacrylate applied topically to the pancreatic stump and anastomosis site during pancreaticojejunostomy. The control group will receive standard duct-to-mucosa pancreaticojejunostomy without adhesive. All patients will receive standardized perioperative care, including prophylactic antibiotics and drain management per ISGPF guidelines.

Follow-up will include daily amylase measurements in drains (days 1,3,5), CT imaging if POPF suspected.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective pancreaticoduodenectomy for malignant lesions.
* Intraoperative confirmation of soft pancreatic texture (by surgeon palpation; friable, non-fibrotic pancreas).
* Age 18-75 years .
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate organ function defined as:

Hemoglobin ≥ 9.0 g/dL Absolute neutrophil count ≥ 1,500/μL Platelet count ≥ 100,000/μL Total bilirubin ≤ 3 times upper limit of normal Alanine transaminase (ALT) /Alanine transaminase (ALT)( ≤ 5 times upper limit of normal Serum creatinine ≤ 1.5 times upper limit of normal

* Informed consent provided.
* Willingness to comply with study procedures and follow-up requirements.

Exclusion Criteria:

* Hard pancreatic texture (intraoperative surgeon assessment).
* Emergency surgery.
* Previous pancreatic surgery or pancreatic anastomosis.
* Intraoperative identification of unresectable disease
* Known allergy to cyanoacrylate or components.
* Pregnancy or lactation.
* Active infection or sepsis.
* Inability to comply with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Pancreatic Fistula (POPF). | 30 days post-surgery.
  Percentage of patients developing postoperative pancreatic fistula as defined by International Study Group on Pancreatic Fistula (ISGPF) criteria. POPF is defined as drain output of any measurable volume of fluid on or after postoperative day 3 with amylase content greater than 3 times the upper normal serum value. Graded as A (biochemical leak), B , or C.

SECONDARY OUTCOMES:
Time to POPF resolution. | 90 days post-surgery.
  Number of days from surgery to complete resolution of pancreatic fistula.
Postoperative complications | 30 days post-surgery
  Incidence of delayed gastric emptying, bile leak, wound infection, intra-abdominal abscess, and other complications.
Reoperation Rate | 90 days post-surgery.
  Percentage of patients requiring reoperation for complications.
Length of Hospital Stay | Up to 90 days
  Total number of days in hospital following surgery(days).
Incidence of postpancreatectomy Hemorrhage | 30 days post-surgery
  Per International Study Group on Pancreatic Fistula (ISGPS) criteria.
Mortality Rate | 90 days post-surgery
  All-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Gaspar AF, Kemp R, Sankarankutty AK, Lopes Junior JR, Filho JAF, Avezum VAPAF, de Assis Mota G, Nunes AA, Dos Santos JS. Influence on Postoperative Results and Cost-effectiveness of Using Cyanoacrylate Glue for Pancreaticojejunal Anastomosis After Duodenopancreatectomy. Pancreas. 2025 Aug 1;54(7):e610-e617. doi: 10.1097/MPA.0000000000002479. PMID 40127250